CLINICAL TRIAL: NCT00584545
Title: Simultaneous Fluoroscopic and Manometric Measures of the Oropharyngeal Phase of Deglutition
Status: Withdrawn | Type: Observational
Why Stopped: Study never got started.
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 200715362
Record Dates: First submitted 2007-12-26; First posted 2008-01-02 (Estimated); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Dysphagia
Keywords: pharyngeal manometry; videofluoroscopy
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To validate the pharyngeal constriction ration, a surrogate measure of pharyngeal strength on fluoroscopy by comparing it with simultaneous pharyngeal manometry.

DETAILED DESCRIPTION:
The specific aim of this study is to validate the pharyngeal constriction ration, a surrogate measure of pharyngeal strength on fluoroscopy by comparing it with simultaneous pharyngeal manometry. Combined videofluoroscopic swallowing studies with pharyngeal manometry are commonly used in the evaluation of dysphagia. However, no published study has compared the results of simultaneous pharyngeal manometry with objective timing and displacement measures on videofluoroscopy. These objective measures, such as the pharyngeal constriction ratio, were developed here at UCD and are not yet routinely used by other practitioners. A secondary aim of this study will be to corroborate recent data in the literature suggesting that the presence of feeding tube through the upper esophageal sphincter does not affect the oropharyngeal phase of deglutition. This topic is currently under hot debate in the speech language pathology realm and has important implications for the evaluation of hospitalized patients with dysphagia.

ELIGIBILITY:
Inclusion Criteria:

* undergone pharyngeal manometry with simultaneous videofluoroscopy during the period 1/1/06 to 4/30/07

Exclusion Criteria:

* those who do not meet the inclusion criteria; pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: UCDMC otolaryngology primary clinic
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Belafsky, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States